CLINICAL TRIAL: NCT02583503
Title: Hindfoot Alignment in TKR - Validation of a Novel Radiographic Study
Brief Title: Hindfoot Alignment in Total Knee Replacement
Status: Completed | Type: Observational
Sponsor: Golden Jubilee National Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: Ortho 15-09
Record Dates: First submitted 2015-09-01; First posted 2015-10-22 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2015-10

CONDITIONS: Osteoarthritis
Keywords: Total knee arthroplasty; Total knee replacement; TKA; TKR
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hindfoot alignment view x ray: Patients undergoing TKR for osteoarthritis will have an additional x ray (hindfoot alignment view) as well as the standard hip knee ankle x ray extended to include the heel.
  Interventions: Radiation: Hindfoot alignment view x ray

INTERVENTIONS:
Radiation: Hindfoot alignment view x ray — Diagnostic x rays used to measure leg alignment.

SUMMARY:
When carrying out a knee replacement operation one of the goals is to correct any deformity of the leg (bowlegged or knock kneed). The ideal alignment is the mechanical axis, which is a line from the centre of the hip joint to the centre of the ankle. This line indicates how the weight of the body is transmitted to the ground via the leg. Often the planning for a knee replacement uses an Xray which shows the hip, knee and ankle (HKA Xray) so that the mechanical axis can be drawn on.

However, the weight of the body goes to the ground from the ankle through the heel. There have been some reports recently suggesting that deformities in the heel can influence the overall leg alignment after a knee replacement; this may affect how successful the surgery is, or how long the knee replacement will last. Therefore it may make sense to take the alignment of the leg including the heel in planning for a knee replacement.

The conventional practice to assess the alignment of the heel is a hindfoot alignment view (HAV) Xray. This only shows the foot. Having two separate Xrays means more radiation exposure and makes linking the two alignments very difficult. We propose a single novel Xray extending the HKA Xray to shows hip, knee, ankle and heel (HKAH Xray) enabling measurement of both alignments.

This study is to validate the hindfoot alignment seen on the novel Xray with the standard HAV. Patients undergoing a knee replacement will be enrolled. Patients will have both a HKAH and HAV Xray before surgery. The alignment of the heel measured on the HKAH Xray will be compared with the standard HAV to see if it is accurate.

DETAILED DESCRIPTION:
Patients going on the waiting list for TKR at our hospital will be enrolled prospectively.

Each patient will have two radiographs preoperatively. One radiograph will be the novel HKAH radiograph to measure the alignment of the heel to the whole leg and the other will be the HAV radiograph which will be used as the standard to which the HKAH measure of alignment will be compared. The HKAH radiograph will be taken instead of the standard care HKA radiograph and the HAV is additional to standard care.

Each participant will receive an information sheet along with the outpatients appointment letter which is dispatched approximately a week in advance of their appointment date. This will carry information about the study, and the risks (one additional radiograph).

Participants who are going to have a knee replacement will have a written & informed consent to take part in the study. If they agree then they will have an additional radiograph before surgery. If they don't agree then they will have a single radiograph before surgery as is the norm in our hospital.

Whether they take part or not will have absolutely no bearing on the treatment they receive, or the aftercare.

ELIGIBILITY:
Inclusion Criteria:

* Predominant knee osteoarthritis requiring total knee replacement
* Able to give informed consent
* Able to return for 6 week follow-up

Exclusion Criteria:

* Advanced osteoarthritis in other lower limb joint(s)
* limb length discrepancy requiring a shoe-raise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients scheduled for a total knee replacement at the Golden Jubilee National Hospital under the care of one of the orthopaedic consultants who have agreed to provide patients for this study.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2015-12-07 (Actual); Primary Completion 2016-06-28 (Actual); Study Completion 2016-06-28 (Actual)

PRIMARY OUTCOMES:
Leg alignment angle measured from the hip knee ankle heel radiograph compared to that measured from the standard hindfoot radiograph. | Baseline
  Leg alignment angle measured from the hip knee ankle heel radiograph compared to that measured from the standard hindfoot radiograph.

CONTACTS AND LOCATIONS:
Overall Officials: Kalpesh Shah, Principal Investigator — Golden Jubilee National Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mullaji A, Shetty GM. Persistent hindfoot valgus causes lateral deviation of weightbearing axis after total knee arthroplasty. Clin Orthop Relat Res. 2011 Apr;469(4):1154-60. doi: 10.1007/s11999-010-1703-z. Epub 2010 Dec 1. PMID 21120711
- [Background] Hara Y, Ikoma K, Arai Y, Ohashi S, Maki M, Kubo T. Alteration of hindfoot alignment after total knee arthroplasty using a novel hindfoot alignment view. J Arthroplasty. 2015 Jan;30(1):126-9. doi: 10.1016/j.arth.2014.07.026. Epub 2014 Jul 25. PMID 25155238